CLINICAL TRIAL: NCT04398745
Title: A Phase I Study to Evaluate the Pharmacokinetics and Safety of Belantamab Mafodotin Monotherapy in Participants With Relapsed and/or Refractory Multiple Myeloma (RRMM) Who Have Normal and Varying Degrees of Impaired Renal Function (DREAMM 12)
Brief Title: A Study of Belantamab Mafodotin Monotherapy in Multiple Myeloma Participants With Normal and Varying Degree of Impaired Renal Function
Acronym: DREAMM12
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209626
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: DREAMM12; End-stage renal disease; Normal renal function; Renal impairment; Relapsed and/or refractory multiple myeloma; Belantamab mafodotin
MeSH Terms: conditions — Multiple Myeloma; Kidney Failure, Chronic; Renal Insufficiency | interventions — belantamab mafodotin

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Participants with normal/mild impaired renal function (Experimental): Participants with normal or mildly impaired renal function (Normal: individual glomerular filtration rate [iGFR]: >=90 milliliter per minute; Mild impairment: iGFR: 60-89 mL/min will be administered with belantamab mafodotin 2.5 mg/kg as an intravenous infusion over 30 minutes Q3W on Day 1 of every 21- day cycle until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, or end of study, whichever occurs first.
  Interventions: Drug: Belantamab mafodotin
- Part 1: Participants with severe renal impairment (Experimental): Participants with severely impaired renal function (iGFR: 15-29 mL/min) will be administered with belantamab mafodotin 2.5 mg/kg as an intravenous infusion over 30 minutes Q3W on Day 1 of every 21- day cycle until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, or end of study, whichever occurs first.
  Interventions: Drug: Belantamab mafodotin
- Part 2: Participants with ESRD (not on dialysis) (Experimental): Participants with ESRD (iGFR: <15 mL/min) not on dialysis will be administered with belantamab mafodotin either 2.5 mg/kg or 1.9 mg/kg (or other adjusted dose) as an intravenous infusion over 30 minutes Q3W on Day 1 of every 21- day cycle until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, or end of study, whichever occurs first. In Part 2, the dose will be decided after evaluation of pharmacokinetic and safety data of Part 1.
  Interventions: Drug: Belantamab mafodotin
- Part 2: Participants with ESRD (on hemodialysis) (Experimental): Participants with ESRD (iGFR: <15 mL/min) on hemodialysis will be administered with belantamab mafodotin either 2.5 mg/kg or 1.9 mg/kg (or other adjusted dose) as an intravenous infusion over 30 minutes Q3W on Day 1 of every 21-day cycle until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, or end of study, whichever occurs first. In Part 2, the dose will be decided after evaluation of pharmacokinetic and safety data of Part 1.
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be provided as lyophilized powder which will be available as 100 milligrams per vial (mg/vial) in single-use vial for reconstitution. Lyophilized belantamab mafodotin will reconstituted using water for injection, dilute with normal 0.9 % saline before use.
  Other Names: GSK2857916

SUMMARY:
Belantamab mafodotin is an antibody-drug conjugate (ADC) containing humanized anti- B-cell maturation antigen (BCMA) monoclonal antibody (mAb). Renal impairment is a major complication of multiple myeloma (MM) and the majority of MM participants is either at risk or already has renal dysfunction at initial diagnosis. The purpose of this study is to assess the pharmacokinetics (PK), safety, and tolerability of belantamab mafodotin monotherapy in participants with RRMM, who have had at least 3 lines of prior treatment (or at least 2 lines of prior treatment if ineligible for autologous stem cell transplantation ) and have either normal or impaired renal functions. The study will consist of two parts: part 1 will include participants with normal/mildly impaired renal function and severe renal impairment and part 2 will include participants with end-stage renal disease (ESRD), where participants are either not undergoing or require hemodialysis. Participants will be administered belantamab mafodotin at a dose of 2.5 milligram per kilogram (mg/kg) intravenously once in three weeks (Q3W) dosing in Part 1. Based on the Part 1 Safety/Pharmacokinetic (PK) data, Part 2 participants will be administered the dose of either 2.5 mg/kg or 1.9 mg/kg (or other adjusted dose). Participants will be treated with belantamab mafodotin monotherapy until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, or end of study, whichever occurs first. This study will include a screening phase, treatment phase, follow-up phase and a post analysis continued treatment (PACT) phase . The total duration of the study is approximately up to 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants are capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the Informed Consent Form.
* Male and/or female participants must be 18 years of age or older, at the time of signing the informed consent. In Republic of Korea, participants must be 19 years of age or older at the time of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Participants with histologically or cytologically confirmed diagnosis of MM, as defined in International Myeloma Working Group criteria: 1. Has undergone autologous stem cell transplant (SCT) or is considered transplant-ineligible; 2. Has failed at least 2 prior lines of anti-myeloma treatments, including an immunomodulatory drug (example [e.g.], lenalidomide or pomalidomide) and a proteasome inhibitor (e.g., bortezomib, ixazomib or carfilzomib). In Republic of Korea, participants should also have relapsed or refractory disease after treatment with an anti-CD38 antibody, if accessible to patients, or other suitable local standard of care.
* Participants have measurable disease with at least one of the following: Serum M-protein >=0.5 grams per deciliter (g/dL) (>=5 grams per liter [g/L]); Urine M-protein >=200 milligrams (mg) per 24 hours (mg/24 h); and Serum free light chain (FLC) assay: Involved FLC level >=10 milligrams per deciliter (mg/dL) (>=100 milligrams per liter [mg/L]) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participants with a history of autologous SCT are eligible for study participation provided the following eligibility criteria are met: 1. Transplant was >100 days prior to study enrollment, 2. No active infection(s), and 3. Participant meets the remainder of the eligibility criteria outlined in this protocol.
* Participants with adequate organ system functions as defined follows: Absolute neutrophil count >=1.0 x 10^9 per liter (/L); Hemoglobin >=7.0 g/dL or 4.9 millimoles per liter (mmol/L); Platelets >= 50 x 10^9/L; Total bilirubin <=1.5 x Upper limit of normal (ULN) (Isolated bilirubin >=1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]); Alanine aminotransferase <=2.5 x ULN; iGFR, Group 1: normal/ mildly impaired >=60milliliter per minute (mL/min); Group 2: severe 15-29 mL/min; Group 3: ESRD (not on dialysis) <15 mL/min; Group 4: ESRD (on dialysis) <15 mL/min; and left ventricular ejection fraction by echocardiograms >=40%.
* Main additional inclusion criteria in Group 1 (matched control participants): Matched to at least one severely renal impaired participant by Baseline body weight (+/-20%) and Baseline albumin levels (+/-10%).
* Female participants: Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) OR is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the intervention period and for at least 4 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. A WOCBP must have a negative highly sensitive serum pregnancy test within 72 hours of dosing on Cycle 1 Day 1 and agree to use highly effective contraception during the study and for 4 months after the last dose of study medication. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Male participants: Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male participants are eligible to participate if they agree to the following from the time of first dose of study until 6 months after the last dose of study treatment to allow for clearance of any altered sperm: Refrain from donating sperm and either; Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; OR must agree to use a male condom even if they have undergone a successful vasectomy and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a WOCBP (including pregnant females).

Exclusion Criteria:

* Participants with active plasma cell leukemia at the time of screening. Symptomatic amyloidosis, active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, myeloma protein and skin changes), Waldenstroem Macroglobulinemia
* Participants had a prior allogeneic stem cell transplant. . Participants who have undergone a syngeneic bone marrow transplant will be allowed only if there is no history of, or no currently active graft-versus-host-diseases (GvHD).
* Participant has received an investigational drug within 14 days or 5 half-lives whichever is shorter, preceding the first dose of study drug. This includes prior treatment with a monoclonal antibody. The only exception is emergency use of a short course of systemic corticosteroids (equivalent to, or less than: dexamethasone 40 milligrams per day [mg/day] for a maximum of 4 days) before treatment.
* Prior belantamab mafodotin therapy.
* Participant has received a strong Organic-anion transporting polypeptide inhibitor within 14 days or 5 half-lives, whichever is shorter, preceding the first dose of study drug.
* Systemic active infection requiring treatment.
* Any unresolved toxicity >=Grade 2 from previous treatment except for alopecia, or peripheral neuropathy up to Grade 2.
* Plasmapheresis within 7 days prior to the first dose of study drug. Screening laboratory values must be performed after last plasmapheresis.
* Any major surgery within the last 4 weeks prior to Day 1 of Screening.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities except renal impairment) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Evidence of active mucosal or internal bleeding.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. (Stable chronic liver disease [(including Gilbert's syndrome or asymptomatic gallstones]) or hepatobiliary involvement of malignancy is acceptable if participant otherwise meets entry criteria)
* Participants with previous or concurrent malignancies other than MM are excluded, unless the prior malignancy has been considered medically stable for at least 2 years. The participant must not be receiving active therapy, other than hormonal therapy for this disease. (Participants with curatively treated non-melanoma skin cancer are allowed without a 2-year restriction)
* Evidence of cardiovascular risk including any of the following: Evidence of current clinically significant untreated arrhythmias, including clinically significant electrocardiogram abnormalities such as second degree (Mobitz Type II) or third degree atrioventricular block; History of myocardial infarction (within prior 18 months), acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening; Class III or IV heart failure as defined by the New York Heart Association functional classification system and uncontrolled hypertension.
* Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
* Known human immunodeficiency virus infection, unless the participant can meet all of the following criteria: Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load <400 copies/mL prior to first dose; CD4+ T-cell (CD4+) counts ≥350 cells/ L and no history of AIDS-defining opportunistic infections within the last 12 months
* Participants with Hepatitis B will be excluded unless the following criteria can be met: If the participant is hepatitis B core antibody (HbcAb) positive or hepatitis B surface antigen (HbsAg) negative, then hepatitis B virus (HBV) deoxyribonucleic acid (DNA) should be undectectable at the time of screening; If HbsAg+ at screening or <=3 months prior to first dose of study treatment, then HBV DNA should be undetectable, highly effective antiviral treatment should be started ≥4 weeks prior to first dose of study treatment. Participants with cirrhosis are excluded.
* Positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid test result at Screening or within 3 months prior to first dose of study treatment unless the participant can meet the following criteria: RNA test negative and Successful anti-viral treatment (usually 8 weeks duration) is required, followed by a negative HCV RNA test after a washout period of at least 4 weeks prior to first dose.
* Participants with renal impairment due to hepatic disease (hepatorenal syndrome).
* Current corneal epithelial disease except for mild punctuate keratopathy.
* Participant is a woman who is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Maximum observed plasma concentration (Cmax) of GSK2857916 | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Time to Cmax (Tmax) of GSK2857916 | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Concentration of GSK2857916 at the end of infusion (C-EOI) | Cycle 1 up to Cycle 3: end infusion (EOI) (each cycle is 21 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Predose plasma concentration (Ctrough) of GSK2857916 | Predose on Cycle 1 and up to Cycle 3 (each cycle is 21 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: AUC over the dosing interval (AUC[0-tau]) of GSK2857916 | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Last time point where the concentration is above the limit of quantification (Tlast) of GSK2857916 | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Cmax of total monoclonal antibody (mAb) | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Tmax of total mAb | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Ctrough of total mAb | Predose on Cycle 1 and up to Cycle 3 (each cycle is 21 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: C-EOI of total mAb | Cycle 1 up to Cycle 3: end infusion (EOI) (each cycle is 21 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: AUC(0-tau) of total mAb | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Tlast of total mAb | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Cmax of Cys Monomethyl Auristatin F (cys-mcMMAF) | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Tmax of cys-mcMMAF | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: C-EOI of cys-mcMMAF | Cycle 1 up to Cycle 3: end infusion (EOI) (each cycle is 21 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: AUC(0-168 hours) of cys-mcMMAF | Predose and up to 168 hours
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 1: Tlast of cys-mcMMAF | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Cmax of GSK2857916 | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Tmax of GSK2857916 | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: C-EOI of GSK2857916 | Cycle 1 up to Cycle 3: end infusion (EOI) (each cycle is 21 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Ctrough of GSK2857916 | Predose on Cycle 1 and up to Cycle 3 (each cycle is 21 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: AUC(0-tau) of GSK2857916 | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Tlast of GSK2857916 | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Cmax of total mAb | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Tmax of total mAb | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: C-EOI of mAb | Cycle 1 up to Cycle 3: end infusion (EOI) (each cycle is 21 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Ctrough of total mAb | Predose on Cycle 1 up to Cycle 3 (each cycle is 21 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: AUC(0-tau) of total mAb | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Tlast of total mAb | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Cmax of cys-mcMMAF | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Tmax of cys-mcMMAF | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: C-EOI of cys-mcMMAF | Cycle 1 up to Cycle 3: end infusion (EOI) (each cycle is 21 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: AUC(0-168 hours) of cys-mcMMAF | Predose and up to 168 hours
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Part 2: Tlast of cys-mcMMAF | Up to Day 85
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.

SECONDARY OUTCOMES:
Part 1 and Part 2: Change from Baseline in Vital Signs- Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) (millimeter of mercury [mmHg]) | Baseline and up to 48 months
  Vital signs will be measured after resting for at least 5 minutes.
Part 1 and Part 2: Change from Baseline in Vital Sign- Heart rate (beats per minute) | Baseline and up to 48 months
  Vital signs will be measured after resting for at least 5 minutes.
Part 1 and Part 2: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 48 months
  AEs and SAEs will be collected at specified time points.
Part 1 and Part 2: Number of participants with toxicity grading for clinical laboratory parameters | Up to 48 months
Part 1 and Part 2: Change from baseline in physical examination parameter | Baseline and up to 48 months
  Physical examination parameter will include assessment of weight only.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (11):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Westwood, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, The Woodlands, Texas
- GSK Investigational Site, Athens, Greece
- GSK Investigational Site, Singapore, Singapore
- South Korea (3):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com